CLINICAL TRIAL: NCT05724602
Title: Radiotherapy Plus Xevinapant or Placebo in Older Patients With Locally Advanced Head and Neck Squamous Cell Carcinoma: a Randomized Phase II Study RAVINA
Brief Title: Radiotherapy Plus Xevinapant in Older Patients With Locally Advanced Head and Neck Squamous Cell Carcinoma
Acronym: RAVINA
Status: Suspended | Phase: Phase 2 | Type: Interventional
Why Stopped: discontinuation of all ongoing studies involving xevinapant
Sponsor: European Organisation for Research and Treatment of Cancer - EORTC (Network)
Collaborators: Merck KGaA, Darmstadt, Germany (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: EORTC 2120-HNCG; EU trial Number (Other: 2022-502339-20-00)
Record Dates: First submitted 2023-01-17; First posted 2023-02-13 (Actual); Last update posted 2024-08-27 (Actual); Status verified 2024-08

CONDITIONS: Locally Advanced Head and Neck Squamous Cell Carcinoma
Keywords: Older adults (≥ 70 years)

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Radiotherapy + Xevinapant (Experimental): 3 cycles of xevinapant (200 mg/day from Day 1 to 14, per 21-day cycle) + IMRT followed by 3 cycles of xevinapant in monotherapy (200 mg/day from Day 1 to 14, per 21-day cycle)
  Interventions: Drug: Xevinapant
- Radiotherapy + Placebo (Placebo Comparator): 3 cycles of placebo (from Day 1 to 14, per 21-day cycle) + IMRT followed by 3 cycles of placebo in monotherapy (from Day 1 to 14, per 21-day cycle).
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: Xevinapant — 3 cycles of xevinapant + IMRT followed by 3 cycles of xevinapant as monotherapy
  Arms: Radiotherapy + Xevinapant
Drug: Placebo — 3 cycles of placebo + IMRT followed by 3 cycles of placebo as monotherapy
  Arms: Radiotherapy + Placebo

SUMMARY:
This is a multicenter, randomized, placebo-controlled, triple blind, phase II study to determine the efficacy and safety of xevinapant with radiotherapy in older patients with locally advanced head and neck squamous cell carcinoma (LA-HNSCC) of oral cavity, oropharynx, hypopharynx, or larynx.

Upon confirmation of eligibility, subjects will be enrolled and randomized in a 1:1 ratio to:

* Arm A: 3 cycles of xevinapant (200 mg/day from Day 1 to 14, per cycle) + intensive modulated radiotherapy (IMRT) followed by 3 cycles of xevinapant in monotherapy phase (200 mg/day from Day 1 to 14, per cycle)
* Arm B: 3 cycles of placebo (from Day 1 to 14, per cycle) + IMRT followed by 3 cycles of placebo in monotherapy phase (from Day 1 to 14, per cycle).

Patients will be stratified by institution, disease location/p16 status (p16 positive oropharyngeal cancer, versus others), G8 score. Three strata for the G8 will be used (>14, versus 11-14 versus <11).

Patients will undergo imaging in week 20 and upon clinical suspicion of progression/recurrence. Clinical examination will take place every 12 weeks in the first 3 years.

ELIGIBILITY:
Main Inclusion Criteria:

* Age ≥ 70 years.
* Pathologically proven new diagnosis of HNSCC of oral cavity, oropharynx, hypopharynx and larynx tumor.
* cT3-4 cN0 cM0 or cT1-4 cN1-3 cM0 except for T1-2N1 p16 positive oropharyngeal cancer (AJCC 8th edition).
* HPV status using p16 immunohistochemistry (IHC) available for oropharyngeal squamous cell carcinoma.
* Measurable disease per RECIST 1.1.
* Eastern Coperative Oncology Group Performance Status (ECOG PS) ≤ 1.
* Intention to treat with curative intent primary radiotherapy alone.
* Able to swallow liquids or has an adequately functioning feeding tube, gastrostomy or jejunostomy placed.
* Adequate hematologic, renal, and hepatic function as indicated by:
* Creatinine clearance ≥ 30 mL/min, measured with the Cockroft and Gault formula.
* Absolute neutrophil count ≥ 1 500 cells/μL.
* Platelets ≥ 100 000 cells/μL.
* Hemoglobin ≥ 9.0 g/dL or ≥5.6 mmol/L (blood transfusions during screening are permitted).
* AST and ALT ≤ 3.0 × upper limit of normal (ULN).
* Total bilirubin ≤ 1.5 × ULN (up to 2.0 × ULN is allowed if the direct bilirubin level is normal and the elevation is limited to indirect bilirubin).
* Written informed consent must be signed according to ICH/GCP, and national/local regulations.

Main Exclusion Criteria:

* Unknown primary, primary nasopharynx and paranasal sinus.
* Two primaries.
* Any previous or current treatment for invasive head and neck cancer, including induction chemotherapy, surgery, concomitant chemotherapy and cetuximab.
* Gastrointestinal disorders that could affect drug absorption.
* Another malignancy in the previous 3 years with exception of curatively treated disease with no evidence of recurrence.
* Known allergy to xevinapant or any excipient known to be present in active or placebo formulation.
* Active gastrointestinal bleeding, or any other uncontrolled bleeding requiring more than 2 red blood cell transfusions or 4 units of packed red blood cells within 4 weeks prior to enrolment
* Non-Decompensated or symptomatic liver cirrhosis (Child-Pugh score: B or C).
* Impaired cardiovascular function or clinically significant cardiovascular diseases
* Any uncontrolled, intercurrent illness or clinical situation that would in the judgment of investigator, limit compliance with study requirements. This includes but is not limited to uncontrolled active infections, defined as any infection requiring IV antibiotics within 7 days prior to enrolment.

Min Age: 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Older Adult
Enrollment: 230 (Estimated)
Dates: Start 2023-11-15 (Actual); Primary Completion 2029-07 (Estimated); Study Completion 2029-10 (Estimated)

PRIMARY OUTCOMES:
Locoregional event-free survival (LREFS) | 5 years after first patient in
  To demonstrate superior efficacy in terms of locoregional event-free survival of xevinapant vs placebo when added to radical radiotherapy in older patients with LA-HNSCC.

SECONDARY OUTCOMES:
Response to treatment by RECIST 1.1 | 5 years after first patient in
  To estimate the added value of xevinapant over RT alone in terms of response to treatment.
Progression Free Survival as assessed by the local investigator | 5 years after first patient in
  To estimate the added value of xevinapant over RT alone in PFS.
Overall Survival | 5 years after first patient in
  To estimate the added value of xevinapant over RT alone in OS.
Safety according to the CTCAE (NCI Common Terminology Criteria for Adverse Events) Version 5.0 for toxicity and Serious Adverse Event reporting | 5 years after first patient in
  To evaluate the frequency and severity of toxicities according to CTCAE v5.0 in the two arms.
HRQOL as assessed by global health/QoL and physical functioning scales at week 20 (Fatigue scale from the Quality of Life Core-30 (QLQ-C30) and pain in the head and neck scale from Item List-225 (IL225)). | 5 years after first patient in
  To assess non-inferiority of xevinapant arm compared to placebo in terms of health-related quality of life (HRQoL) as assessed by the EORTC QLQ-C30 global health/QoL and physical functioning scales.
  The questionnaires employ 50 4-point Likert scales with responses from "not at all" to "very much" and two 7-point Likert scales for global health and overall HRQoL. For functional and global HRQoL scales, higher scores represent a better level of functioning and are converted to a 0 to 100 scale. For symptom-oriented scales, a higher score represents more severe symptoms.

CONTACTS AND LOCATIONS:
Overall Officials: Sjoukje Oosting, Dr, Study Chair — University Medical Center Groningen; Pierluigi Bonomo, Dr, Study Chair — Azienda Ospedaliero-Universitaria Careggi
Locations (26):
- Belgium (3):
  - Onze Lieve Vrouw Ziekenhuis, Aalst
  - Universitair Ziekenhuis Gent, Ghent
  - Cliniques Universitaires Saint-Luc, Woluwe-Saint-Lambert
- France (4):
  - Centre Oscar Lambret, Lille
  - Institut de Cancerologie de Lorraine, Nancy
  - Assistance Publique Hopitaux Paris- APHP - APHP Sorbonne Univ - Hopital la Pitie-Salpetriere, Paris
  - Assistance Publique Hopitaux Paris- APHP - APHP Sorbonne Univ - Hopital Tenon, Paris
- Germany (3):
  - Charite - Universitaetsmedizin Berlin - Campus Virchow-Klinikum, Berlin
  - Universitaetsklinikum - Essen, Essen
  - Universitaets Krankenhaus Eppendorf - Universitaetsklinikum Hamburg-Eppendorf KE - University Cancer Center, Hamburg
- Ireland (2):
  - University Hospital Galway, Galway
  - St Luke Hospital & SLRON - SLRON - St. Luke'S Hospital Rathgar, Rathgar
- Italy (3):
  - IRCCS--Ospedale Bellaria-Bologna, Bologna
  - Univ. of Florence -Azienda Ospedaliero-Universitaria Careggi, Florence
  - Istituto Clinico Humanitas, Rozzano
- Netherlands (3):
  - Amsterdam UMC - locatie VUMC, Amsterdam
  - Universitair Medisch Centrum Groningen - University Medical Center Groningen, Groningen
  - Academisch Ziekenhuis Maastricht, Maastricht
- Norway (2):
  - Helse Bergen HF -Haukeland Hospital - Univ. Hosp, Bergen
  - Oslo University Hospital - Radiumhospitalet, Oslo
- The Institute Of Oncology, Ljubljana, Slovenia
- Spain (2):
  - Institut Catala d'Oncologia - ICO L'Hospitalet - Hospital Duran i Reynals, Barcelona
  - Vall D Hebron - Hospital Universitari Vall d'Hebron, Barcelona
- United Kingdom (3):
  - The Clatterbridge cancer Center NHS foundation Trust - Clatterbridge Cancer Center - Wirral, Birkenhead
  - University Hospitals Bristol NHS Foundation Trust - Bristol Haematology And Oncology Centre, Bristol
  - NHS Greater Glasgow and Clyde - Beatson West of Scotland Cancer Centre - Gartnavel General Hospital, Glasgow